CLINICAL TRIAL: NCT05233085
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Doses of AZD4041 in Healthy Adult Subjects
Brief Title: A Safety Study of AZD4041 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Altasciences Company Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7460C00002; UG3DA054825 (NIH); NCT05209334 (obsolete NCT alias)
Record Dates: First submitted 2021-12-14; First posted 2022-02-10 (Actual); Results first posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Opioid Use Disorder (OUD)
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: For each cohort, 9 participants will be randomly assigned to receive AZD4041 and 3 participants will be assigned to receive placebo. Within each cohort, 2 participants will be randomized initially to AZD4041 or placebo (1:1 ratio) to allow a sentinel dosing approach. Providing no clinically significant issues have been noted after the first 3 doses of the initial 2 (sentinel) participants in a cohort and provided the Day 3 safety laboratory tests for the 2 participants have been reviewed, the remaining 10 participants will be randomized to AZD4041 or placebo in an 8:2 ratio. All participants will receive either AZD4041 or placebo administered once daily for 14 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: AZD4041 Dose Level 1 (Experimental): Participants will receive oral solution of AZD4041 dose level 1 once daily (QD) directly into the mouth using a syringe from Days 1 to 14.
  Interventions: Drug: AZD4041
- Cohort 2: AZD4041 Dose Level 2 (Experimental): Participants will receive oral solution of AZD4041 dose level 2 QD directly into the mouth using a syringe from Days 1 to 14.
  Interventions: Drug: AZD4041
- Cohort 3: AZD4041 Dose Level 3 (Experimental): Participants will receive oral solution of AZD4041 dose level 3 QD directly into the mouth using a syringe from Days 1 to 14.
  Interventions: Drug: AZD4041
- Cohorts 1-3: Pooled Placebo (Placebo Comparator): Participants will receive oral solution of placebo equivalent to AZD4041 volume QD directly into the mouth using a syringe from Days 1 to 14.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD4041 — Participants will receive oral solution of AZD4041 as stated in arm description.
  Arms: Cohort 1: AZD4041 Dose Level 1; Cohort 2: AZD4041 Dose Level 2; Cohort 3: AZD4041 Dose Level 3
Other: Placebo — Participants will receive oral solution of placebo as stated in arm description.
  Arms: Cohorts 1-3: Pooled Placebo

SUMMARY:
This is a Phase 1, single-centre, randomized, double-blind, placebo-controlled, multiple ascending doses (MAD) study in healthy male and female adult participants.

The study will include up to 48 participants (12 participants per cohort) who will be randomized 9:3 to active drug or placebo. Each cohort will receive AZD4041 or placebo in a MAD study.

A sequential cohort MAD design will be employed to assure that higher doses are administered to healthy participants only after lower doses have demonstrated an acceptable safety profile.

The total study duration will be up to 59 days (including Screening) per participant.

ELIGIBILITY:
Inclusion Criteria

* Provision of signed and dated written informed consent form prior to any study specific procedures
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Healthy adult male or female participants. Female participants must be of non-childbearing potential (postmenopausal and/or surgically sterile)
* If female, meets one of the following criteria:

  1. Physiological postmenopausal status, defined as the following:

     1. absence of menses for at least 12 months following cessation of all exogenous hormonal treatments (without an alternative medical condition) at Screening and prior to the first study drug administration; and
     2. follicle stimulating hormone (FSH) levels ≥ 40 mIU/mL at Screening; and
     3. must have a negative pregnancy test result at screening and check-in. and/or
  2. Surgical sterile, defined as those who have had:

hysterectomy, bilateral oophorectomy and/or bilateral salpingectomy, or bilateral tubal ligation. Women who are surgically sterile must provide documentation of the procedure by an operative report, ultrasound, or other verifiable documentation; and must have a negative pregnancy test result at screening and check-in.

If postmenopausal and has an FSH of < 40 mIU/mL, but meets all other criteria in (1) or (2) above as well as all the other inclusion criteria, screening oestradiol serum level must be equal to or below 150 pmol/L.

* Men who are biologically capable of fathering children must agree and commit to use an adequate form of contraception for the duration of the treatment period and for no less than 120 days (4 months) after the last administration of study intervention. A male participant is considered capable of fathering children even if his sexual partner is sterile or using contraceptives.
* Men who are biologically capable of fathering children must also agree to refrain from sperm donation for the duration of the treatment period and for at least 90 days after the last administration of study intervention.
* Aged at least 18 years but not older than 55 years on the day of randomization
* Body mass index (BMI) within 18.0 kg/m^2 to 30.0 kg/m^2, inclusive
* Body weight of within 50 kg to 100 kg, inclusive
* Non- or ex-smoker (An ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration)
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical or neurological examination (including vital signs) and/or ECG and/or safety laboratory tests, as determined by an Investigator
* Suitable veins for cannulation or repeated venepuncture

Exclusion Criteria

* Female who is lactating
* Female who is pregnant according to the pregnancy test at Screening or prior to the first study drug administration
* Male participants with a history of oligospermia or azoospermia or any other disorder of the reproductive system
* Male participants who are undergoing treatment or evaluation for infertility.
* History of significant allergy/ hypersensitivity to AZD4041 or products related to AZD4041 as well as severe allergy/hypersensitivity reactions (like angioedema) to any drugs
* Presence or history of significant gastrointestinal, liver or kidney disease, or any other condition that is known to interfere with drug absorption, distribution, metabolism, or excretion, or known to potentiate or predispose to undesired effects
* History of any significant disease, including [but not necessarily limited to] significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, or dermatologic disease
* Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 21 units/week or > 3 units/day for men; > 14 units/week or > 2 units/day for women; intake of excessive alcohol, acute or chronic)
* History of any significant psychiatric disorder according to the criteria of the Diagnostic and Statistical manual of Mental Disorders, 5th Edition (DSM-5, American Psychiatric Association 2013) which, in the opinion of the Investigator, could be detrimental to participant safety or could compromise study data interpretation.
* History of substance use disorder, other than nicotine or caffeine (as per DSM-5 criteria)
* Use of any prescription drugs, including hormone replacement therapy in the 28 days prior to the first study drug administration, that in the opinion of an Investigator would put into question the status of the participant as healthy
* Use of St. John's wort in the 28 days prior to the first study drug administration
* Positive test result for alcohol and/or drugs of abuse at Screening or prior to the first study drug administration
* Any clinically significant illness, medical/surgical procedure or trauma within the 28 days prior to the first study drug administration
* Any abnormal or clinically significant findings in laboratory test results at Screening that would, in the opinion of an Investigator, increase the participant's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data
* Positive screening results to human immunodeficiency virus (HIV) antigen/antibody (Ag/Ab) combo, hepatitis B surface antigen, or hepatitis C virus tests
* Showing suicidal tendency as per the C-SSRS questionnaire administered at Screening
* Any abnormal vital signs, after 10 minutes supine rest, as defined in the list below, at the Screening Visit/or Day -2 Out of range tests may be repeated once for each visit at the discretion of an Investigator.

  1. Systolic blood pressure (BP) < 90 mmHg or >140 mmHg
  2. Diastolic BP < 50 mmHg or > 90 mmHg
  3. Heart Rate < 45 or > 85 beats per minute (bpm)
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG which, in an Investigator's opinion, may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol-defined primary lead or left ventricular hypertrophy at Screening or prior to the first study drug administration
* Prolonged QT interval corrected for HR using Fridericia's formula (QTcF) > 440 ms at Screening or prior to the first study drug administration
* Shortened QTcF < 340 ms at Screening or prior to first study drug administration
* Known family history of long QT syndrome
* ECG interval measured from the onset of the P wave to the onset of the complex between Q and S waves (QRS complex) (PR [PQ]) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular preexcitation) at Screening or prior to the first study drug administration
* PR (PQ) interval prolongation (> 220 ms), persistent or intermittent second (Wenckebach block while asleep is not exclusive), or third degree atrioventricular (AV) block, or AV dissociation at Screening or prior to the first study drug administration
* Persistent or intermittent complete bundle branch block, incomplete bundle branch block, or intraventricular conduction delay (IVCD) with ECG interval measured from the onset of the QRS complex to the J point (QRS) > 110 ms. Participants with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of ventricular hypertrophy or preexcitation at Screening or prior to the first study drug administration
* In the pre-dose 24 hour telemetry, presence of ≥ 10 ventricular premature contractions (VPCs) during 1 hour, or ≥ 100 VPCs during 24-hours of telemetry, or any occurrence of paired VPC (ventricular couplets) or other repetitive ventricular rhythms, including non-sustained or sustained (> 30 second duration), slow (< 100 bpm), or fast (≥ 100 bpm) ventricular tachycardias.
* Vaccination with the Coronavirus disease 2019 (COVID-19) vaccine less than 14 days prior to first study dose administration
* Scheduled immunization with a COVID-19 vaccine (first or second dose) during the study that, in the opinion of an Investigator, could potentially interfere with participant participation, participant safety, study results, or any other reason
* Use of any prescribed or nonprescribed oral and topical inhibitors/inducers of CYP3A4 (including shampoo).
* Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) as judged by an Investigator
* Participants who have previously received AZD4041
* Any history of tuberculosis
* Involvement of any AstraZeneca or study site employee or their close relatives
* Judgment by an Investigator that the participant should not participate in the study if they have any ongoing or recent (ie, during the Screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements
* Presence of any tongue piercings or history of any tongue piercings in the last 90 days prior to the first study drug administration
* Participants who have medical dietary restrictions
* Participants who cannot communicate reliably with the Investigator
* Inclusion in a previous group for this clinical study
* Intake of an investigational product (IP) within at least 28 days or 5 half-lives; whichever is longer, prior to the first study drug administration
* Donation of 50 mL or more of blood in the 28 days prior to the first study drug administration
* Donation of 500 mL or more of blood in the 56 days prior to the first study drug administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Laval, Quebec, Canada

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7460C00002&attachmentIdentifier=2e3c7ff6-0213-4cd6-b3cc-56996b032ecf&fileName=azd4041-d7460c00002-synopsis_Redacted.pdf&versionIdentifier=
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7460C00002&attachmentIdentifier=72c5b28a-78bc-4784-8966-f286d88db443&fileName=D7460C00002-Statistical_Analysis_Plan_Redacted.pdf&versionIdentifier=
- See also: Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7460C00002&attachmentIdentifier=e33e69e8-6900-49cc-90aa-1e51c7d31dfe&fileName=D7460C00002-Protocol_Amendment_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: AZD4041 Dose Level 1: Participants received oral solution of AZD4041 dose level 1 once daily (QD) directly into the mouth using a syringe from Days 1 to 14.
- Cohort 2: AZD4041 Dose Level 2: Participants received oral solution of AZD4041 dose level 2 QD directly into the mouth using a syringe from Days 1 to 14.
- Cohort 3: AZD4041 Dose Level 3: Participants received oral solution of AZD4041 dose level 3 QD directly into the mouth using a syringe from Days 1 to 14.
- Cohorts 1-3: Pooled Placebo: Participants received oral solution of placebo equivalent to AZD4041 volume QD directly into the mouth using a syringe from Days 1 to 14.
Period: Overall Study
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3 | Cohorts 1-3: Pooled Placebo
Started | 9 | 9 | 9 | 9
Completed | 8 | 9 | 9 | 9
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of AZD4041 or placebo.
Groups:
- Cohort 1: AZD4041 Dose Level 1: Participants received oral solution of AZD4041 dose level 1 QD directly into the mouth using a syringe from Days 1 to 14.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3 | Cohorts 1-3: Pooled Placebo | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.9 (11.7) | 37.1 (8.9) | 40.2 (10.8) | 41.6 (11.6) | 40.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 1
  Male | 9 | 9 | 9 | 8 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 5 | 0 | 12
  Not Hispanic or Latino | 5 | 6 | 4 | 9 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 8 | 8 | 8 | 8 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: From Day 1 to Day 31
Population: Safety population included all participants who received at least 1 dose of AZD4041 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3 | Cohorts 1-3: Pooled Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Any TEAEs | 8 | 6 | 6 | 9
  Any TESAEs | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormal finding in the vital sign parameters (blood pressure, pulse rate, and body temperature).
Time Frame: From Day 1 to Day 31
Population: Safety population included all participants who received at least 1 dose of AZD4041 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3 | Cohorts 1-3: Pooled Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 1 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs
Description: Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported. Abnormal clinical laboratory parameters defined as any abnormal finding during analysis of general biochemistry, hematology, and urinalysis.
Time Frame: From Day 1 to Day 31
Population: Safety population included all participants who received at least 1 dose of AZD4041 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3 | Cohorts 1-3: Pooled Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal Electrocardiograms (ECGs) Reported as TEAEs
Description: Number of participants with abnormal ECGs reported as TEAEs are reported.
Time Frame: From Day 1 to Day 31
Population: Safety population included all participants who received at least 1 dose of AZD4041 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3 | Cohorts 1-3: Pooled Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Ventricular tachycardia | 1 | 0 | 1 | 1
  Sinus tachycardia | 1 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Suicidal Ideation or Behavior Assessed Using Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is described as a scale developed at Columbia University that has 2-6 questions each in categories of Suicidal Ideation, Intensity of Ideation, Suicidal Behavior, and Actual Attempts. Four constructs were measured. Severity of Suicidal ideation is rated on a 5-point ordinal scale. Intensity of ideation is comprised of 5 items (frequency, duration, controllability, deterrents, and reason for ideation), each rated on a 5-point ordinal scale. Suicidal behavior is rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and non-suicidal self-injurious behavior. Lethality, assesses actual attempts; actual lethality is rated on a 6-point ordinal scale, and if actual lethality is 0, potential lethality of attempts is rated on a 3-point ordinal scale.The higher the C-SSRS score, the higher the suicide risk (ie. worse outcome).
Time Frame: Baseline (Days -28 to -1) through Day 17
Population: Safety population included all participants who received at least 1 dose of AZD4041 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3 | Cohorts 1-3: Pooled Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Suicidal ideation | 0 | 0 | 0 | 0
  Suicidal behavior | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Clinically Significant Findings in Physical and Neurological Examinations
Description: Number of participants with clinically significant findings in physical and neurological examinations are reported.
Time Frame: Baseline (Days -28 to -1) through Day 31
Population: Safety population included all participants who received at least 1 dose of AZD4041 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3 | Cohorts 1-3: Pooled Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Abnormal Male Hormone Levels as Assessed by the Investigator
Description: Male hormone levels investigated included testosterone, luteinizing hormone, follicle stimulating hormone, and inhibin B. Number of Participants with abnormal male hormone levels as assessed by the investigator are reported.
Time Frame: Day -1, pre-dose and 1.5 hours post-dose on Days 1 and 14
Population: Safety population included all participants who received at least 1 dose of AZD4041 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3 | Cohorts 1-3: Pooled Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of AZD4041 After Day 1 Dose
Description: The Cmax of AZD4041 after Day 1 dose is reported.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours postdose
Population: Pharmacokinetic (PK) population included all participants who had received at least 1 dose of AZD4041 and had at least 1 PK concentration after dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 9 | 9 | 9
ng/mL | 165.93 (24.3) | 377.85 (25.7) | 590.78 (12.6)

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of AZD4041 After Day 14 Dose
Description: The Cmax of AZD4041 after Day 14 dose is reported.
Time Frame: Day 14: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: Pharmacokinetic (PK) population included all participants who had received at least 1 dose of AZD4041 and had at least 1 PK concentration after dosing. Here, number of participants analyzed (N) indicates those participants who had adequate PK samples and excludes participants with inadequate PK samples due to missed blood draw, an AE, meal deviation, or concomitant medication intake.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 8 | 9 | 9
ng/mL | 232.44 (20.7) | 478.10 (21.7) | 940.99 (25.7)

10. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of AZD4041 After Day 1 Dose
Description: The Tmax of AZD4041 after Day 1 dose is reported.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours postdose
Population: The PK population included all participants who had received at least 1 dose of AZD4041 and had at least 1 PK concentration after dosing.
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 9 | 9 | 9
Hour | 1.05 [0.50 to 1.53] | 1.00 [0.25 to 1.50] | 1.02 [0.55 to 1.50]

11. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of AZD4041 After Day 14 Dose
Description: The Tmax of AZD4041 after Day 14 dose is reported.
Time Frame: Day 14: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: The PK population included all participants who had received at least 1 dose of AZD4041 and had at least 1 PK concentration after dosing. Here, number of participants analyzed (N) indicates those participants who had adequate PK samples and excludes participants with inadequate PK samples due to missed blood draw, an AE, meal deviation, or concomitant medication intake.
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 8 | 9 | 9
Hour | 1.02 [0.50 to 2.00] | 1.02 [0.50 to 1.52] | 1.00 [0.50 to 3.02]

12. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 24 Hours (AUC0-24) of AZD4041 After Day 1 Dose
Description: The AUC0-24 of AZD4041 after Day 1 dose is reported.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours postdose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 9 | 9 | 9
h*ng/mL | 1802.21 (21.4) | 3682.61 (25.2) | 6951.39 (20.1)

13. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 (Dose Administration) to the Time of Last Quantifiable Concentration (AUC0-t) of AZD4041 After Day 1 Dose
Description: The AUC0-t of AZD4041 after Day 1 dose is reported.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours postdose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 9 | 9 | 9
h*ng/mL | 1802.90 (21.4) | 3683.15 (25.2) | 6953.42 (20.1)

14. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 (Dose Administration) to the Time of Last Quantifiable Concentration (AUC0-t) of AZD4041 After Day 14 Dose
Description: The AUC0-t of AZD4041 after Day 14 dose is reported.
Time Frame: Day 14: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 8 | 9 | 9
h*ng/mL | 4808.19 (60.1) | 9573.98 (47.0) | 20969.29 (49.6)

15. Secondary Outcome: Area Under the Concentration-time Curve Extrapolated to Infinity (AUC0-inf) of AZD4041 After Day 1 Dose
Description: The AUC0-inf of AZD4041 after Day 1 dose is reported. This PK parameter (AUC0-inf) requiring apparent elimination rate constant (λz) estimation was not evaluable for Cohorts 1 and 3 due to meeting either the exclusion criteria R^2 < 0.8 or the extrapolated area > 20%.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours postdose
Population: as for outcome 11
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 0 | 1 | 0
h*ng/mL |  | 3000.93 [3000.93 to 3000.93] |

16. Secondary Outcome: Area Under the Concentration-time Curve Over the Dosing Interval at Steady State (AUCτ) of AZD4041 After Day 14 Dose
Description: The AUCτ of AZD4041 calculated after Day 14 dose is reported.
Time Frame: Day 14: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 8 | 9 | 9
h*ng/mL | 3022.57 (41.3) | 6306.52 (34.4) | 12622.32 (36.0)

17. Secondary Outcome: Observed Concentration at the End of the Dosing Interval (Ctrough) of AZD4041
Description: The Ctrough of AZD4041 is reported.
Time Frame: Predose on Days 2 (Day 1, 24-hours), 3, 4, 5, 6, 7, 8, 9, 10, 14
Population: The PK population included all participants who had received at least 1 dose of AZD4041 and had at least 1 PK concentration after dosing. Here, number analyzed (n) denotes those participants who were analyzed for the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 9 | 9 | 9
ng/mL
  Day 2 | 45.5 (39.2) | 86.2 (45.2) | 193 (35.2)
  Day 3: number analyzed (Participants) | 8 | 9 | 9
  Day 3 | 62.5 (46.9) | 113 (48.9) | 285 (39.4)
  Day 4: number analyzed (Participants) | 8 | 9 | 9
  Day 4 | 64.9 (52.4) | 124 (56.2) | 314 (43.9)
  Day 5: number analyzed (Participants) | 8 | 9 | 9
  Day 5 | 65.4 (54.6) | 134 (48.4) | 317 (46.2)
  Day 6: number analyzed (Participants) | 8 | 9 | 9
  Day 6 | 69.3 (63.6) | 139 (56.5) | 336 (46.5)
  Day 7: number analyzed (Participants) | 8 | 9 | 9
  Day 7 | 68.4 (64.8) | 141 (55.2) | 331 (45.8)
  Day 8: number analyzed (Participants) | 8 | 9 | 9
  Day 8 | 73.2 (55.6) | 158 (53.6) | 359 (44.4)
  Day 9: number analyzed (Participants) | 8 | 9 | 9
  Day 9 | 73.3 (59.1) | 152 (61.6) | 349 (49.9)
  Day 10: number analyzed (Participants) | 8 | 9 | 9
  Day 10 | 75.0 (62.8) | 158 (62.9) | 341 (46.9)
  Day 14: number analyzed (Participants) | 8 | 9 | 9
  Day 14 | 82.0 (64.6) | 164 (70.8) | 371 (51.9)

18. Secondary Outcome: Concentration at the End of the Dosing Interval (Cτ) of AZD4041 After Day 14 Dose
Description: The Cτ of AZD4041 after Day 14 dose is reported.
Time Frame: Day 14: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 8 | 9 | 9
ng/mL | 81.23 (63.2) | 168.42 (62.0) | 358.37 (56.5)

19. Secondary Outcome: Terminal Elimination Half-life (t1/2,z) of AZD4041 After Day 1 Dose
Description: The t1/2,z of AZD4041 after Day 1 dose is reported. This PK parameter (t1/2,z) requiring λz estimation was not evaluable for Cohorts 1 and 3 due to meeting either the exclusion criteria R^2 < 0.8 or the extrapolated area > 20%.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours postdose
Population: as for outcome 11
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 0 | 1 | 0
hour |  | 8.30 [8.30 to 8.30] |

20. Secondary Outcome: Terminal Elimination Half-life (t1/2,z) of AZD4041 After Day 14 Dose
Description: The t1/2,z of AZD4041 after Day 14 dose is reported.
Time Frame: Day 14: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 6 | 9 | 7
Hour | 18.87 (27.5) | 20.07 (33.4) | 23.22 (20.3)

21. Secondary Outcome: Effective Half-life (t1/2Eff) of AZD4041 After Day 14 Dose
Description: The t1/2Eff of AZD4041 after Day 14 dose is reported.
Time Frame: Day 14: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 8 | 9 | 9
Hour | 17.02 (50.9) | 18.35 (38.7) | 20.33 (34.2)

22. Secondary Outcome: Accumulation Ratio Evaluated by Comparing Day 14 Cmax to Day 1 Cmax (RAC[Cmax]) of AZD4041
Description: The RAC(Cmax) of AZD4041 is reported.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours postdose; Day 14: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 8 | 9 | 9
Ratio | 1.38 (20.9) | 1.27 (22.4) | 1.59 (16.0)

23. Secondary Outcome: Accumulation Ratio Evaluated by Comparing Day 14 AUCτ to Day 1 AUC0-24 (RAC[AUC]) of AZD4041
Description: The RAC(AUC) of AZD4041 is reported.
Time Frame: as for outcome 22
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 8 | 9 | 9
Ratio | 1.66 (25.3) | 1.71 (21.7) | 1.82 (22.1)

24. Secondary Outcome: Apparent Total Clearance (CL/F) of AZD4041 After Day 1 Dose
Description: The CL/F of AZD4041 after Day 1 dose is reported. This PK parameter (CL/F) requiring λz estimation was not evaluable for Cohorts 1 and 3 due to meeting either the exclusion criteria R^2 < 0.8 or the extrapolated area > 20%.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours postdose
Population: as for outcome 11
Measure: Median (Full Range); unit: L/hour
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 0 | 1 | 0
L/hour |  | 5.00 [5.00 to 5.00] |

25. Secondary Outcome: Apparent Total Clearance at Steady State (CL/Fss) of AZD4041 After Day 14 Dose
Description: The CL/Fss of AZD4041 after Day 14 dose is reported.
Time Frame: Day 14: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 8 | 9 | 9
L/hour | 2.48 (41.3) | 2.38 (34.4) | 1.98 (36.0)

26. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of AZD4041 After Day 1 Dose
Description: The Vz/F of AZD4041 after Day 1 dose is reported. This PK parameter (Vz/F) requiring λz estimation was not evaluable for Cohorts 1 and 3 due to meeting either the exclusion criteria R^2 < 0.8 or the extrapolated area > 20%.
Time Frame: Day 1: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours postdose
Population: as for outcome 11
Measure: Median (Full Range); unit: L
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 0 | 1 | 0
L |  | 59.90 [59.90 to 59.90] |

27. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vz/Fss) of AZD4041 After Day 14 Dose
Description: The Vz/Fss of AZD4041 after Day 14 dose is reported.
Time Frame: Day 14: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 8 | 9 | 9
L | 79.50 (21.8) | 68.90 (25.5) | 75.90 (16.0)

28. Secondary Outcome: Apparent Elimination Rate Constant (λZ) of AZD4041 After Day 14 Dose
Description: The λZ of AZD4041 after Day 14 dose is reported.
Time Frame: Day 14: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 6 | 9 | 7
1/hour | 0.0367 (27.5) | 0.0345 (33.4) | 0.0298 (20.3)

29. Secondary Outcome: Amount of AZD4041 Excreted Unchanged in Urine Over the 24-hour Dosing Interval (Ae0-24) After Day 1 Dose
Description: The Ae0-24 of AZD4041 after Day 1 dose is reported.
Time Frame: Day 1: Predose spot collection, and 0 to 6 hours, 6 to 12 hours, and 12 to 24 hours postdose
Population: The PK population included all participants who had received at least 1 dose of AZD4041 and had at least 1 PK concentration after dosing. Here, number of participants analyzed (N) indicates those participants who had adequate urine PK samples and excludes participants with inadequate urine PK samples due to missed urine collection, an AE, meal deviation, or concomitant medication intake.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 8 | 9 | 8
ng | 59209.58 (71.1) | 161067.17 (71.1) | 411420.17 (45.7)

30. Secondary Outcome: Amount of AZD4041 Excreted Unchanged in Urine Over the 24-hour Dosing Interval (Ae0-24) After Day 14 Dose
Description: The Ae0-24 of AZD4041 after Day 14 dose is reported.
Time Frame: Day 14: Predose spot collection, and 0 to 6 hours, 6 to 12 hours, and 12 to 24 hours postdose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 6 | 8 | 8
ng | 177681.47 (55.3) | 334754.86 (99.2) | 1095233.64 (39.7)

31. Secondary Outcome: Apparent Fraction of AZD4041 Excreted Unchanged in Urine Over the 24-hours Dosing Interval (fe/F0-24) After Day 1 Dose
Description: The fe/F0-24 of AZD4041 after Day 1 dose is reported.
Time Frame: Day 1: Predose spot collection, and 0 to 6 hours, 6 to 12 hours, and 12 to 24 hours postdose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 8 | 9 | 8
Percentage | 0.79 (71.1) | 1.07 (71.1) | 1.65 (45.7)

32. Secondary Outcome: Apparent Fraction of AZD4041 Excreted Unchanged in Urine Over the 24-hours Dosing Interval (fe/F0-24) After Day 14 Dose
Description: The fe/F0-24 of AZD4041 after Day 14 dose is reported.
Time Frame: Day 14: Predose spot collection, and 0 to 6 hours, 6 to 12 hours, and 12 to 24 hours postdose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 6 | 8 | 8
Percentage | 2.37 (55.3) | 2.23 (99.2) | 4.38 (39.7)

33. Secondary Outcome: Apparent Renal Clearance Over the 24-hours Dosing Interval (CLR 0-24) of AZD4041 After Day 1 Dose
Description: The CLR 0-24 of AZD4041 after Day 1 dose is reported. Apparent renal clearance was calculated as: Ae (0-24) / AUC0-24 on Day 1.
Time Frame: Day 1: Predose spot collection, and 0 to 6 hours, 6 to 12 hours, and 12 to 24 hours postdose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 8 | 9 | 8
L/hour | 0.0328 (65.3) | 0.0437 (72.1) | 0.0582 (56.1)

34. Secondary Outcome: Apparent Renal Clearance Over the 24-hours Dosing Interval (CLR 0-24) of AZD4041 After Day 14 Dose
Description: The CLR 0-24 of AZD4041 after Day 14 dose is reported. Apparent renal clearance was calculated as: Ae (0-24) / AUCτ on Day 14.
Time Frame: Day 14: Predose spot collection, and 0 to 6 hours, 6 to 12 hours, and 12 to 24 hours postdose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 6 | 8 | 8
L/hour | 0.0536 (21.5) | 0.0521 (106.4) | 0.0916 (71.2)

35. Secondary Outcome: Cerebrospinal Fluid (CSF) Concentration as a Percentage of Total Plasma Concentration of AZD4041 in Cohorts 2 and 3
Description: The CSF concentration as a percentage of total plasma concentration of AZD4041 in cohorts 2 and 3 is reported.
Time Frame: Day 14 post dose (approximately 3 hours ± 1 hour)
Population: The PK population included all participants who had received at least 1 dose of AZD4041 and had at least 1 PK concentration after dosing. Here, number of participants analyzed (N) indicates those participants who had adequate CSF PK samples and excludes participants with inadequate CSF PK samples due to missed CSF draw, an AE, meal deviation, or concomitant medication intake.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 6 | 9
Percentage | 4.91 (13.3) | 5.28 (16.3)

36. Secondary Outcome: CSF Concentration as a Percentage of Free Plasma Concentration of AZD4041 in Cohorts 2 and 3
Description: The CSF concentration as a percentage of free plasma concentration of AZD4041 in cohorts 2 and 3 is reported.
Time Frame: Day 14 post dose (approximately 3 hours ± 1 hour)
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3
Number analyzed (Participants) | 6 | 9
Percentage | 27.44 (13.3) | 29.51 (16.3)

37. Secondary Outcome: Day 14 / Day 1 Ratio of 4-β-hydroxy-cholesterol Concentrations
Description: Day 14 / Day 1 ratio of 4-β-hydroxy-cholesterol concentrations is reported.
Time Frame: Pre-dose Day 1 and 24 hours post Day 14 dose
Population: Pharmacodynamic (PD) population included all participants who had received at least 1 dose of AZD4041 or placebo and had at least 1 plasma 4-β-hydroxy-cholesterol concentration after dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3 | Cohorts 1-3: Pooled Placebo
Number analyzed (Participants) | 8 | 9 | 9 | 9
Ratio | 1.00 (28.67) | 1.02 (18.83) | 0.95 (18.74) | 0.79 (26.41)

ADVERSE EVENTS:
Time Frame: From Day 1 to Day 31
Description: Safety population included all participants who received at least 1 dose of AZD4041 or placebo.
Arm/Group | Cohort 1: AZD4041 Dose Level 1 | Cohort 2: AZD4041 Dose Level 2 | Cohort 3: AZD4041 Dose Level 3 | Cohorts 1-3: Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 8/9 | 6/9 | 6/9 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: AZD4041 Dose Level 1 (N=9) | Cohort 2: AZD4041 Dose Level 2 (N=9) | Cohort 3: AZD4041 Dose Level 3 (N=9) | Cohorts 1-3: Pooled Placebo (N=9)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site reaction (General disorders) | 6 (9) | 0 (0) | 3 (5) | 6 (12)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 3 (9) | 3 (11)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (5) | 2 (2) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT05233085/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT05233085/SAP_001.pdf